CLINICAL TRIAL: NCT01899105
Title: A Phase 1, Randomized, Single-Dose, Open-Label Crossover Study to Investigate the Effect of Food on the Relative Bioavailability of 2 Fixed-Dose Combinations of Lumacaftor and Ivacaftor Tablet Formulations in Healthy Adult Subjects
Brief Title: A Phase 1 Study to Investigate the Food Effect of Lumacaftor in Combination With Ivacaftor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: VX13-809-012
Record Dates: First submitted 2013-07-10; First posted 2013-07-15 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor; ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): A single dose of 2 fixed-dose combination tablets of 200mg lumacaftor/125mg ivacaftor (total of 400mg lumacaftor/250mg ivacaftor) in the fed state and fasted state with a 14 day washout period in between each dosing occasion
  Interventions: Drug: lumacaftor; Drug: ivacaftor
- Part B (Experimental): A single dose of 3 fixed-dose combination tablets of 200mg lumacaftor/83mg ivacaftor (total of 600mg lumacaftor and 250mg ivacaftor) in the fed with a 14 day washout period in between dosing occasions
  Interventions: Drug: lumacaftor; Drug: ivacaftor

INTERVENTIONS:
Drug: lumacaftor
  Other Names: VX-809
Drug: ivacaftor
  Other Names: VX-770

SUMMARY:
This study is designed to investigate the effect of food on the relative bioavailability of 2 different strengths of fixed-dose combinations of lumacaftor and ivacaftor tablet formulations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects as defined in the protocol
* Subjects who weigh >50 kg at Screening

Exclusion Criteria:

* History of any illness or condition that might confound the results of the study or pose an additional risk to the subject upon administration of study drug - Positive for hepatitis B,C, or HIV
* Standard 12-lead ECG demonstrating QTc >450 msec for male subjects and >480 msec for female subjects at the Screening Visit
* Abnormal renal function as defined in the protocol at Screening
* Forced expiratory volume in 1 second (FEV1) <80% predicted at the Screening Visit
* Blood donation (of approximately 1 pint [500 mL] or more) within 56 days before the first dose of study drug
* Treatment with an investigational drug or device within 30 days or 5 half-lives preceding the first dose of study drug

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of lumacaftor and ivacaftor, including Cmax, AUC0-tlast, and AUC0-∞ | up to 5 days

SECONDARY OUTCOMES:
Safety and tolerability as assessed by adverse events (AEs), laboratory assessments (serum chemistry and hematology), vital signs, standard 12-lead electrocardiograms (ECGs), and spirometry | up to 25 days

CONTACTS AND LOCATIONS:
Locations (1):
- Daytona Beach, Florida, United States

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662